CLINICAL TRIAL: NCT02423642
Title: Immunomodulation Effect of Regional Citrate Anticoagulation in Acute Kidney Injury Requiring Continuous Renal Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Division of Nephrology, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB.136/56
Record Dates: First submitted 2015-03-31; First posted 2015-04-22 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury Requiring Continuous Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy; Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AKI requring CRRT and use regional citrate anticoagulation (Experimental): CRRT use regional citrate anticoagulation
  Interventions: Procedure: Continuous renal replacement therapy with regional citrate anticoagulation
- AKI requring CRRT and not use regional citrate anticoagulation (Experimental): CRRT not use regional citrate anticoagulation
  Interventions: Procedure: Continuous renal replacement therapy with no anticoagulation or heparin

INTERVENTIONS:
Procedure: Continuous renal replacement therapy with regional citrate anticoagulation — CRRT with anticoagulant : regional citrate anticoagulation
  Filter : AQUAMAX™ (Edwards Lifesciences)
  Other Names: Continuous veno-venous hemofiltration
  Arms: AKI requring CRRT and use regional citrate anticoagulation
Procedure: Continuous renal replacement therapy with no anticoagulation or heparin — CRRT with any anticoagulant : no anticoagulation or heparin Filter : AQUAMAX™ (Edwards Lifesciences)
  Other Names: Continuous veno-venous hemofiltration
  Arms: AKI requring CRRT and not use regional citrate anticoagulation

SUMMARY:
The purpose of this study is to study the effect of anticoagulation in immune response with Acute Kidney Injury (AKI) undergoing Continuous Renal Replacement Therapy (CRRT).

ELIGIBILITY:
Inclusion Criteria:

* Systemic inflammatory response syndrome; SIRS > or = 2 meets definition
* Patients with acute kidney injury in the intensive care ward.
* Requiring continuous renal replacement therapy.

Exclusion Criteria:

* Pregnancy
* Cirrhosis
* End stage renal disease
* HIV infection
* Serum creatinine in male > 2 mg/dl and female > 1.5 mg/dl
* Bleeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Functions of inflammatory cells | 24 hours
  CD11b expression on PMN and HLA-DR expression on monocyte
Regulation of inflammatory reactions and and opsonization in microorganisms | 24 hours
  C3a and C5a
Activity of acute phase protein during acute inflammation | 24 hours
  PAI-1

SECONDARY OUTCOMES:
survival rate | 28 days
length of ICU stay | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sasipha Tachaboon, Bangkok, Pathumwan, Thailand

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078